CLINICAL TRIAL: NCT01318057
Title: Pharmacogenetics of Warfarin in Puerto Rican Patients Using a Physiogenomics Approach.
Brief Title: Pharmacogenetics of Warfarin in Puerto Ricans.
Status: Completed | Type: Observational
Sponsor: University of Puerto Rico (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Hartford Hospital (Other); VA Caribbean Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jorge Duconge, PhD, MSc, BSc Pharm, Professor, University of Puerto Rico
Other Study IDs: 1SC2HL110393-01A2 (NIH); SC2HL110393 (NIH)
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Atrial Fibrillation; Deep Vein Thrombosis; Cardiac Valvular Insufficiency; Antiphospholipid Syndrome; Coagulopathy
Keywords: Pharmacogenetics; Warfarin; Personalized Medicine; Puerto Ricans; Physiogenomics; Hispanics; Anticoagulants; Cardiovascular; Deep Vein Thrombosis with or without Pulmonary Embolism; Cardiac Valvular Replacement
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Antiphospholipid Syndrome; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole fresh blood and Genomic DNA samples fom enrolled patients
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Wild-Type: Wild-Type are those individuals who were non-carriers of any functional (loss-of-function)variant in CYP2C9 and/or VKORC1 genes
- Carriers: Those patients who were identified as having any functional CYP2C9 and/or VKORC1 polymorphism

SUMMARY:
Warfarin (Coumadin) is a prescribed "blood thinner" medication used to make the blood less thick in people with high risk of forming blood clots. Despite the various methods to monitor this drug, life-threatening bleeding is a common undesired effect and might result in patient death. Patients starting warfarin therapy may require several weeks or even months to reach the appropriate blood level of warfarin. This blind practice could place the patient at high risk. There are several demographic and clinical factors that significantly influence how much warfarin the patient needs to attain the desired response. Genes, which control hereditary traits, are also important. Now, the investigators know that by using the information encoded in patient's genes the investigators are able to individualize the therapy. Two genes are considered to be involved in warfarin response (CYP2C9 and VKORC1). This study proposes to ascertain what CYP2C9 and VKORC1 variants are present in warfarin-treated Puerto Rican patients. To this purpose, a novel physiogenomic array comprising 384 variants in 222 genes of cardio-metabolic relevance will be used so the investigators are able to determine the structure of the Puerto Rican population in terms of ancestral contributions and how the admixture may impact the prevalence of CYP2C9 and VKORC1 variants. Secondly, the investigators will assess the association of these variants to clinical responses in order to develop a better method of dose estimation. The expected result is the improvement of warfarin therapy in Puerto Ricans. The proposed study will fill a gap in the knowledge of warfarin pharmacogenetics, providing new information on the prevalence of CYP2C9 (metabolism) and VKORC1 (sensitivity) polymorphisms in Puerto Ricans as well as their role in the warfarin response variability observed in this admixed population.

DETAILED DESCRIPTION:
Warfarin is a frequently prescribed drug for both the treatment and prevention of thromboembolic complications. Although many reports have been published over the past years in different populations worldwide, there is a fundamental gap in understanding whether variations in CYP2C9 and VKORC1 genes account for the inter-individual variability in response to warfarin that is observed in Puerto Rican patients. This study is a first step toward the development of DNA-driven personalized guidelines for warfarin dose optimization in Puerto Rican patients with thromboembolic complications. Guided by strong preliminary data, this application will pursuit two specific aims: 1) Develop a physiogenomic (PG)-driven admixture analysis of 350 samples from a population of warfarin-treated Puerto Rican patients using the PG array in order to study the pharmacogenetics of warfarin in Puerto Ricans and 2) Determine whether combinatorial CYP2C9 and VKORC1 genotypes are associated with clinical phenotypes during warfarin therapy in Puerto Rican patients. Under the first aim, 350 DNA specimens from warfarin-treated Puerto Rican patients who consent to participate in this study will be genotyped at large-scale using a novel Illumina-based PG-array of 222 candidate genes from relevant cardio-metabolic and neuro-endocrine pathways in order to examine the population structure of Puerto Ricans and create a reference database of individual admixture, allele frequencies, linkage disequilibrium (LD) and haplotypes for pharmacogenetics studies. Noteworthy, this information remains to be determined in Puerto Ricans. Under the second aim, demographic and clinically relevant non-genetic data will be retrospectively collected from medical records of these patients in order to perform an association analysis between their previously obtained CYP2C9 and VKORC1 genotypes and the corresponding time to achieve stable warfarin dosing following survival analysis techniques and Cox proportional hazards model. Accomplishment of this specific aim will also give the basis for developing a DNA-guided warfarin dosing algorithm in Puerto Rican by using these patients as a learning sample. The long-term goal is to generate valuable information from the genetic background of Puerto Ricans in order to further validate the pharmacogenetic-driven warfarin dosing algorithm for this admixed population. The proposed research is significant because it is expected to advance and expand understanding of how these clinically relevant variants affect the way people from an admixed, under-served population respond to warfarin. This is an important and under-investigated area of pharmacogenetics in minority populations that will have potential applicability to personalize warfarin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose parents are both Puerto Ricans; male and female aged > 18 years old
* Scheduled to receive the standard 5 mg/day oral dose of warfarin for therapeutic anti-coagulation in indications such as deep vein thrombosis (DVT) with or without Pulmonary Embolism (PE)
* Atrial fibrillation (AF) or other arrhythmias, cardiac valvular replacement, and previously diagnosed coagulopathy
* Hematocrit (Hct) > 40%
* Blood Urea Nitrogen (BUN)/creatinine < 30/1.5 mg/dL
* Patients having the ability to understand the requirements of the study and to comply with study procedures and protocol
* Female patient is eligible to enter the study if she is of child-bearing potential but not pregnant or nursing, or not of child-bearing potential

Exclusion Criteria:

* Patients currently enrolled in another active research protocol at the Veteran Affairs Caribbean Healthcare System (VACHS) Hospital
* Blood Urea Nitrogen (BUN)/creatinine > 30/2.0 mg/dL
* Active hepatic disease (defined by a Child-Pugh score above 10 points)
* Ascites
* Total bilirubin above 2.0 mg/dl
* Serum albumin below 3.5 g/dl
* Prothrombin time in seconds prolonged over control > 4
* Hepatic encephalopathy
* Prolonged diarrhea (three or more days)
* Nasogastric or enteral feedings
* Acute illness (e.g., sepsis, infection, anemia)
* Lymphocyte function test (LFT)> 3x upper limit of normal (ULN)
* Active malignancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hispanic Puerto Rican patients from all geographic regions of the Island of Puerto Rico who are currently receiving a standard stable dose of warfarin at the anticoagulation clinic of the Veteran Affair Caribbean Healthcare System (VACHS)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2011-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
time to achieve stable warfarin dose | 6 months
  time to get a stable warfarin dose is defined by the time span (days) from the initial dose until achieving three consecutive INR measurements within therapeutic range (2-3 or 2.5-3.5, according to indication.

SECONDARY OUTCOMES:
time to first bleeding | 6 months
  time to first bleeding is defined as the time span (days) from the initiation of therapy until the first report of serious or life-threatening bleeding episode.
time to first INR>4 | 6 months
  time to first INR above 4 is an indicator of overanticoagulation that is defined as the time span (days) from the initiation of therapy until the first measurement of INR above 4.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle T Rivera-Miranda, PharmD, Principal Investigator — VACHS at San Juan; Jorge Duconge, PhD, Principal Investigator — University of Puerto Rico
Locations (1):
- Veteran Affair Caribbean Healthcare System, San Juan, Puerto Rico

REFERENCES:
- [Background] Villagra D, Duconge J, Windemuth A, Cadilla CL, Kocherla M, Gorowski K, Bogaard K, Renta JY, Cruz IA, Mirabal S, Seip RL, Ruano G. CYP2C9 and VKORC1 genotypes in Puerto Ricans: A case for admixture-matching in clinical pharmacogenetic studies. Clin Chim Acta. 2010 Sep 6;411(17-18):1306-11. doi: 10.1016/j.cca.2010.05.021. Epub 2010 May 19. PMID 20488169
- [Background] Seip RL, Duconge J, Ruano G. Implementing genotype-guided antithrombotic therapy. Future Cardiol. 2010 May;6(3):409-24. doi: 10.2217/fca.10.6. PMID 20462345
- [Background] Duconge J, Cadilla CL, Windemuth A, Kocherla M, Gorowski K, Seip RL, Bogaard K, Renta JY, Piovanetti P, D'Agostino D, Santiago-Borrero PJ, Ruano G. For the patient. DNA makeup of Hispanic persons should be determined before warfarin prescription. Ethn Dis. 2009 Autumn;19(4):479-80. No abstract available. PMID 20077595
- [Background] Duconge J, Cadilla CL, Windemuth A, Kocherla M, Gorowski K, Seip RL, Bogaard K, Renta JY, Piovanetti P, D'Agostino D, Santiago-Borrero PJ, Ruano G. Prevalence of combinatorial CYP2C9 and VKORC1 genotypes in Puerto Ricans: implications for warfarin management in Hispanics. Ethn Dis. 2009 Autumn;19(4):390-5. PMID 20073138
- [Background] Ruano G, Duconge J, Windemuth A, Cadilla CL, Kocherla M, Villagra D, Renta J, Holford T, Santiago-Borrero PJ. Physiogenomic analysis of the Puerto Rican population. Pharmacogenomics. 2009 Apr;10(4):565-77. doi: 10.2217/pgs.09.5. PMID 19374515
- [Background] Rodriguez-Velez R, Ortiz-Rivera OJ, Bower B, Gorowski K, Windemuth A, Villagra D, Kocherla M, Seip RL, D'Agostino D, Vergara C, Ruano G, Duconge J. Exposure to non-therapeutic INR in a high risk cardiovascular patient: potential hazard reduction with genotype-guided warfarin (Coumadin) dosing. P R Health Sci J. 2010 Dec;29(4):402-8. PMID 21261182
- [Background] Duconge J, Ruano G. The Emerging Role of Admixture in the Pharmacogenetics of Puerto Rican Hispanics. J Pharmacogenomics Pharmacoproteomics. 2010 Oct 4;1(101):1000101. doi: 10.4172/2153-0645.1000101. PMID 23227441
- [Background] Duconge J, Cadilla CL. CYP2D6's functional status associated with the length of hospitalization stay in psychiatric patients: a twist in the tale or evidence that matters? Biomark Med. 2013 Dec;7(6):913-4. doi: 10.2217/bmm.13.109. No abstract available. PMID 24266824
- [Result] Ramos AS, Seip RL, Rivera-Miranda G, Felici-Giovanini ME, Garcia-Berdecia R, Alejandro-Cowan Y, Kocherla M, Cruz I, Feliu JF, Cadilla CL, Renta JY, Gorowski K, Vergara C, Ruano G, Duconge J. Development of a pharmacogenetic-guided warfarin dosing algorithm for Puerto Rican patients. Pharmacogenomics. 2012 Dec;13(16):1937-50. doi: 10.2217/pgs.12.171. PMID 23215886
- [Result] Valentin II, Vazquez J, Rivera-Miranda G, Seip RL, Velez M, Kocherla M, Bogaard K, Cruz-Gonzalez I, Cadilla CL, Renta JY, Feliu JF, Ramos AS, Alejandro-Cowan Y, Gorowski K, Ruano G, Duconge J. Prediction of warfarin dose reductions in Puerto Rican patients, based on combinatorial CYP2C9 and VKORC1 genotypes. Ann Pharmacother. 2012 Feb;46(2):208-18. doi: 10.1345/aph.1Q190. Epub 2012 Jan 24. PMID 22274142
- [Result] Orengo-Mercado C, Nieves B, Lopez L, Valles-Ortiz N, Renta JY, Santiago-Borrero PJ, Cadilla CL, Duconge J. Frequencies of Functional Polymorphisms in Three Pharmacokinetic Genes of Clinical Interest within the Admixed Puerto Rican Population. J Pharmacogenomics Pharmacoproteomics. 2013 Mar 27;4(113):1000113. doi: 10.4172/2153-0645.1000113. PMID 24040574
- [Result] Valentin II, Rivera G, Nieves-Plaza M, Cruz I, Renta JY, Cadilla CL, Feliu JF, Seip RL, Ruano G, Duconge J. Pharmacogenetic association study of warfarin safety endpoints in Puerto Ricans. P R Health Sci J. 2014 Sep;33(3):97-104. PMID 25244877
- [Derived] Duconge J, Ramos AS, Claudio-Campos K, Rivera-Miranda G, Bermudez-Bosch L, Renta JY, Cadilla CL, Cruz I, Feliu JF, Vergara C, Ruano G. A Novel Admixture-Based Pharmacogenetic Approach to Refine Warfarin Dosing in Caribbean Hispanics. PLoS One. 2016 Jan 8;11(1):e0145480. doi: 10.1371/journal.pone.0145480. eCollection 2016. PMID 26745506